CLINICAL TRIAL: NCT00324987
Title: A Phase III Randomized Study of Imatinib, With or Without Bevacizumab (NSC-704865), in Patients With Metastatic or Unresectable Gastrointestinal Stromal Tumors
Brief Title: Imatinib Mesylate With or Without Bevacizumab in Treating Patients With Metastatic or Unresectable Gastrointestinal Stromal Tumor
Acronym: S0502
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial failed to accrue
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00776; NCI-2009-00776 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000482236; S0502 (Other: SWOG); S0502 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Results first posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-08

CONDITIONS: Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (CLOSED TO ACCRUAL 10/1/2009) (imatinib and bevacizumab) (Experimental): Patients receive imatinib mesylate PO QD on days 1-21 and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Imatinib Mesylate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm II (CLOSED TO ACCRUAL 10/1/2009) (imatinib) (Active Comparator): Patients receive imatinib mesylate PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Imatinib Mesylate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
  Arms: Arm I (CLOSED TO ACCRUAL 10/1/2009) (imatinib and bevacizumab)
Drug: Imatinib Mesylate — Given PO
  Other Names: CGP 57148; CGP57148B; Gleevec; Glivec; STI 571; STI-571; STI571
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This randomized phase III trial studies imatinib mesylate and bevacizumab to see how well they work compared to imatinib mesylate alone in treating patients with gastrointestinal stromal tumor that has spread to other parts of the body or cannot be removed by surgery. Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. It is not yet known whether imatinib mesylate and bevacizumab are more effective than imatinib mesylate alone in treating gastrointestinal stromal tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether treatment with imatinib (imatinib mesylate) plus bevacizumab leads to improved progression free survival (PFS) versus treatment with imatinib alone in first-line treatment of incurable gastrointestinal stromal tumor (GIST).

SECONDARY OBJECTIVES:

I. To compare response probabilities (confirmed and unconfirmed complete response [CR] and partial response [PR] for subset of patients with measurable disease), overall survival, and central-review based progression-free survival (CRb-PFS) in patients treated with imatinib and bevacizumab versus those treated with imatinib alone.

II. To compare the frequency and severity of toxicities associated with imatinib plus bevacizumab versus imatinib alone.

TERTIARY OBJECTIVES:

I. To explore the association between soluble vascular endothelial growth factor (VEGF), VEGF-factor D (VEGF-D), VEGF receptor (VEGFR)-1, VEGFR-2, angiopoietin-2 (Ang-2), platelet-derived growth factor receptor (PDGFR)-AA and PDGFR-BB levels, positron emission tomography (PET) imaging and immunohistochemistry for cyclin-dependent kinase inhibitor 2A (p16), VEGF and VEGFR, with kinase mutation status and clinical outcomes.

II. To explore imatinib pharmacokinetics with single nucleotide polymorphisms involving the adenosine triphosphate (ATP)-binding cassette, sub-family G (WHITE), member 2 (ABCG2) and cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) genes, as well as other genes that are reported to influence the absorption, distribution, metabolism and elimination of imatinib.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I (CLOSED TO ACCRUAL 10/1/2009): Patients receive imatinib mesylate orally (PO) once daily (QD) on days 1-21 and bevacizumab intravenously (IV) over 30-90 minutes on day 1.

ARM II (CLOSED TO ACCRUAL 10/1/2009): Patients receive imatinib mesylate PO QD on days 1-21.

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 1 month, every 6 months for 2 years, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION # 1
* Patient must have a biopsy proven diagnosis of gastrointestinal stromal tumor (GIST) that is distantly metastatic or unresectable; patients must be determined to be unresectable for cure
* Patient may have measurable and/or non-measurable disease; computed tomography (CT) or magnetic resonance imaging (MRI) used for measurable disease must have been completed within 28 days prior to registration; CT or MRI used for non-measurable disease must have been completed within 42 days prior to registration; PET scans are not sufficient for disease assessment; all disease must be assessed and documented on the Baseline Tumor Assessment Form
* CT/MRI scans must be performed and submitted for central review; archived tissue must be submitted as outlined
* Institutions must seek additional patient consent for PET scans as outlined; if patient consents to the submission of PET scans, the patient must also be registered to Registration #2
* Patient must not have known brain metastasis
* Patient must have a Zubrod performance status of 0 - 3
* Patient must have resolution of transient toxicities from any prior chemotherapy, radiation therapy or surgery to =< grade 1 (Common Terminology Criteria for Adverse Events [CTCAE] version 3.0)
* Patient may have previously received traditional chemotherapeutic agents in any setting, provided at least 28 days have elapsed since completing chemotherapy and they have recovered to =< grade 1 from all drug-induced toxicities
* Patient must not have received prior treatment with bevacizumab or other agents targeting VEGF, VEGFR, or PDGFR for advanced disease; those agents may have been used in the adjuvant setting if the patient did not recur for at least 12 months following the completion of treatment; patients may be receiving imatinib for advanced disease prior to registration provided they meet ALL of the following criteria:

  * Patient must not have received more than 30 days of imatinib treatment prior to registration
  * Patients have not been restaged; (baseline disease assessments prior to initiation of imatinib must fulfill requirements)
  * Patients must have no clinical signs of progression
* Prior radiotherapy is allowed, provided at least 28 days have elapsed since the last treatment and there is evidence of progressive disease within the radiation field or disease outside the radiation field
* Patient must not have had a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration, or anticipation of need for major surgical procedure during the course of the study; no fine needle aspirations or core biopsies are allowed within 7 days prior to registration; no procedure to place a port-a-cath is allowed within 7 days prior to registration
* Patient must have a total bilirubin =< 2.0 x institutional upper limit of normal (IULN), obtained within 28 days prior to registration
* Patients without liver involvement must have serum glutamic oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) =< 2.5 x IULN, obtained within 28 days prior to registration; patients with liver involvement must have SGOT or SGPT =< 5 x IULN
* Patient must have adequate renal function as defined by a serum creatinine =< 1.5 x IULN obtained within 28 days prior to registration
* Patient must have urine protein/creatinine ratio (UPC) < 1; this result must be obtained within 28 days prior to registration
* Patient must have an absolute neutrophil count (ANC) >= 1,000/mcl obtained within 28 days prior to registration
* Patient must have a platelet count >= 100,000/mcl obtained within 28 days prior to registration
* Patient must have hemoglobin >= 9 gm/dl (this may be achieved by transfusion if needed) obtained within 28 days prior to registration
* Patient must have an international normalized ratio (INR) =< 1.5, obtained within 28 days prior to registration
* Patient must have a partial thromboplastin time (PTT) =< IULN, obtained within 28 days prior to registration
* Patient must not be taking therapeutic doses of Coumadin (warfarin) as anticoagulation at the time of registration; patients requiring therapeutic anticoagulation may use low-molecular weight heparin (e.g., Lovenox) or other agents, and mini-dose Coumadin (1 mg PO QD) as prophylaxis is allowed
* Patient must not have had a cerebrovascular accident (CVA), transient ischemic attack (TIA), myocardial infarction or unstable angina within 6 months prior to registration; patient must not have serious cardiac arrhythmia requiring medication, New York Heart Association (NYHA) class II or greater congestive heart failure, or clinically significant peripheral vascular disease
* Patient must not have had an abdominal fistula, gastrointestinal perforation or intraabdominal abscess within 28 days prior to registration
* Patient must not plan to use other investigational agents while on protocol treatment
* Patient must have no contraindication to oral medications (e.g., severe dysphagia); patients with gastrostomy (G)- or jejunostomy (J)- tubes are eligible
* Patient must not have blood pressure > 160/90; patients with a history of hypertension must be on a stable regimen of anti-hypertensive therapy
* Patient must not have a serious, non-healing wound, ulcer, or bone fracture
* Patient must not be pregnant or nursing; male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout protocol treatment and for up to 6 months following discontinuation of study drugs
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* If day 28 or 42 falls on a weekend or holiday, the limit may be extended to the next working day; in calculating days of tests and measurements, the day a test or measurement is done is considered day 0; therefore, if a test is done on a Monday, the Monday four weeks later would be considered day 28
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and identification (ID) number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base
* REGISTRATION #2 - PET SUBSTUDY:
* Patient must have been registered to the main study
* Patient must have consented to the submission of PET scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Blanke, Principal Investigator — SWOG Cancer Research Network
Locations (192):
- United States (190):
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - Marin General Hospital, Greenbrae, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Sutter Cancer Research Consortium, Novato, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - John B Amos Cancer Center, Columbus, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Rush - Copley Medical Center, Aurora, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Adventist La Grange Memorial Hospital, La Grange, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Franciscan St. Francis Health-Beech Grove, Beech Grove, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - Highland Hospital, Rochester, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Adventist Medical Center, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Geisinger South Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Audie L Murphy Veterans Affairs Hospital, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Group Health Cooperative of Puget Sound Oncology Consortium, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (2):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia

REFERENCES:
- [Derived] Blanke CD, Rankin C, Corless C, Eary JF, Mulder K, Okuno SH, George S, Heinrich M. S0502: A SWOG Phase III Randomized Study of Imatinib, With or Without Bevacizumab, in Patients With Untreated Metastatic or Unresectable Gastrointestinal Stromal Tumors. Oncologist. 2015 Dec;20(12):1353-4. doi: 10.1634/theoncologist.2015-0295. Epub 2015 Nov 17. PMID 26576593

RESULTS

PARTICIPANT FLOW:
Groups:
- Imatinib + Bevacizumab: Patients receive 400 or 800mg imatinib mesylate PO QD on days 1-21 and 15 mg/kg bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
- Imatinib: Patients receive 400 or 800mg imatinib mesylate PO QD on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Imatinib + Bevacizumab | Imatinib
Started | 6 | 6
Completed | 0 (Patients were to be treated until progression) | 0 (Patients were to be treated until progression)
Not Completed | 6 | 6
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Progression | 1 | 1
Not completed — symptomatic deterioration, toxicity, etc | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib + Bevacizumab | Imatinib | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Median (Full Range); unit: years] | 64.7 [49.4 to 82.9] | 57.9 [44.0 to 68.5] | 59.9 [44.0 to 82.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Performance Status [Number; unit: participants] — Patients graded according to the Zubrod Perfromance Status Scale:
  0: Fully active, able to carry on all pre-disease performance without restriction; 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light sedentary nature; 2: Ambulatory and capable of self-care but unable to carry out any work activities, up and about more than 50% of waking hours; 3: Capable of limited self-care, confined to bed or chair more than 50% of waking hours; 4: Completely disabled, cannot carry on any self-care, totally confined to bed or chair.
  participants
    0 | 5 | 4 | 9
    >=1 | 1 | 2 | 3
Disease Status [Number; unit: participants]
  Measurable | 5 | 5 | 10
  Non-measurable | 1 | 1 | 2

OUTCOME MEASURES:

1. Secondary Outcome: Response Rate
Description: Confirmed response (CR) is two or more objective statuses of CR a minimum of four weeks apart documented before progression or symptomatic deterioration. Partial response (PR) is two or more objective statuses of PR or better a minimum of four weeks apart documented before progression or symptomatic deterioration. Unconfirmed CR is one objective status of CR documented before progression or symptomatic deterioration but not qualifying as CR or PR. Unconfirmed PR is one objective status of PR documented before progression or symptomatic deterioration but not qualifying as CR, PR or unconfirmed CR.
Time Frame: Up to 7 years
Population: Only eligible and evaluable patients included. No scientific conclusions were forthcoming because of the small number of patients entered in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Imatinib + Bevacizumab | Imatinib
Number analyzed (Participants) | 3 | 5
Participants
  Unconfirmed CR | 0 | 1
  Stable/No Response | 1 | 2
  Assessment Inadequate | 2 | 2

2. Primary Outcome: Progression Free Survival
Description: From date of registration (defined as date of randomization) to date of first observation of progressive disease, death due to any cause or symptomatic deterioration. Patients last known to be alive and progression free are censored at last date of contact. Progression is defined as one or more of the following: 20% increase in the sum of longest diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy), provided at least one target lesion does NOT demonstrate uniform hypoattenuation over > 90% of maximal cross sectional area; unequivocal progression of non-measurable disease; appearance of new lesion/site that is not uniformly hypoattenuating; a hyperattenuating region within a previously cystic/uniformly hypoattenuating lesion will be considered progressive disease if hyperattenuating region is either >= 1 cm in longest diameter or round/oval and forms acute margins with border of target lesion; death due to disease.
Time Frame: Up to 7 years
Population: No scientific conclusions were forthcoming because of the small number of patients entered in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imatinib + Bevacizumab | Imatinib
Number analyzed (Participants) | 6 | 6
months | 30 [8 to 62] | 81 [13 to 81]

3. Secondary Outcome: Overall Survival
Description: From date of registration (defined as date of randomization) to date of death due to any cause. Patients last known to be alive are censored at last date of contact. Note: median was not reached in the Imatinib arm due to limited follow-up data.
Time Frame: up to 7 years
Population: No scientific conclusions were forthcoming because of the small number of patients entered in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imatinib + Bevacizumab | Imatinib
Number analyzed (Participants) | 6 | 6
months | 30 [16 to 30] | 0 [15 to 0]

4. Secondary Outcome: Central-review Based Progression-free Survival (CRb-PFS)
Description: From date of registration (defined as date of randomization) to date of first documentation of one of the following events: death; first documentation of progression based on central review of the appropriate computed tomography (CT) or magnetic resonance imaging (MRI) scans; development of new lesions or disease not identified on CT or MRI; or symptomatic deterioration. Patients not experiencing any of these events will be censored at last date of contact.
Time Frame: up to 7 years
Population: Data not collected as study accrued only 2% of the 572 patients planned. No scientific conclusions were forthcoming because of the small number of patients entered in the study.
Arm/Group | Imatinib + Bevacizumab | Imatinib
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 7 years
Population: Eligible patients who received any treatment and were assessed for adverse events are included in this summary.
Measure: Number; unit: Participants
Arm/Group | Imatinib + Bevacizumab | Imatinib
Number analyzed (Participants) | 5 | 6
Participants
  Fatigue (asthenia, lethargy, malaise) | 1 | 0
  Hemoglobin | 1 | 0
  Hemorrhage, GI - Upper GI NOS | 1 | 0
  INR (of prothrombin time) | 0 | 1
  Proteinuria | 1 | 0
  Thrombosis/embolism (vascular access-related) | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 7 years
Description: Eligible patients who received any treatment and were assessed for adverse events are included in the adverse event summaries.
Arm/Group | Imatinib + Bevacizumab | Imatinib
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/6
Other Adverse Events (participants affected / at risk) | 2/5 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib + Bevacizumab (N=5) | Imatinib (N=6)
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib + Bevacizumab (N=5) | Imatinib (N=6)
Hemoglobin (Blood and lymphatic system disorders) | 2 | 2
Palpitations (Cardiac disorders) | 0 | 1
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 | 0
Vision-blurred vision (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Hemorrhage, GI - Stomach (Gastrointestinal disorders) | 0 | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Edema: head and neck (General disorders) | 0 | 1
Edema: limb (General disorders) | 1 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 | 2
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 0 | 1
Rigors/chills (General disorders) | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Sinus (Infections and infestations) | 1 | 0
Bruising (in absence of Gr 3-4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 | 0
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 1 | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 | 1
AST, SGOT (Investigations) | 1 | 1
Creatinine (Investigations) | 1 | 1
INR (of prothrombin time) (Investigations) | 0 | 1
Leukocytes (total WBC) (Investigations) | 0 | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 | 1
Weight gain (Investigations) | 0 | 1
Weight loss (Investigations) | 1 | 0
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 0 | 1
Pain - Head/headache (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hemorrhage, Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
Trial was terminated due to poor accrual. No conclusions should be drawn from the reported data due to the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less